CLINICAL TRIAL: NCT05201391
Title: Examining the Feasibility and Acceptability of an App-based Mindfulness Intervention for Sexual Minority Women With a History of Early Life Adversities (ELA): A Single Arm Trial
Brief Title: An App-based Mindfulness Intervention for Sexual Minority Women With a History of Early Life Adversities (ELA)
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Brown University (Other)
Collaborators: National Institute on Aging (NIA) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: #2106003013; R24AG065174 (NIH)
Record Dates: First submitted 2021-11-24; First posted 2022-01-21 (Actual); Last update posted 2022-07-08 (Actual); Status verified 2022-07

CONDITIONS: Overweight and Obesity
Keywords: mindfulness-based intervention; weight management; sexual and gender minorities; adverse childhood experiences; mobile application
MeSH Terms: conditions — Overweight; Obesity; Coitus

STUDY DESIGN:
Intervention Model Description: "Eat Right Now" (ERN) is an app-based (28 daily modules, self-paced) Mindfulness-Based Intervention (MBI), which uses mindfulness to target craving-based eating. The program is designed to take 6-8 weeks to complete.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- "Eat Right Now" (ERN) mobile application (Experimental): Participants in this single-arm trial will receive the ERN app as the intervention.
  Interventions: Behavioral: "Eat Right Now" (ERN) mobile application

INTERVENTIONS:
Behavioral: "Eat Right Now" (ERN) mobile application — "Eat Right Now" (ERN) is an app-based (28 daily modules, self-paced) Mindfulness-Based Intervention (MBI), which uses mindfulness to target craving-based eating. The program is designed to take 6-8 weeks to complete.

SUMMARY:
Sexual minority women (SMW) in mid-age are at significantly higher risk for obesity, which is associated with greater vulnerability to cardiovascular disease, diabetes, cancer, and mortality. Further, this group also has elevated risk of early life adversities (ELA), such as childhood trauma and abuse. ELA has been linked to increased risks of midlife obesity and food addiction. However, interventions addressing this public health issue among SMW is scarce. Mindfulness-based interventions (MBI), delivered via smartphone, could be an effective approach to reduce the dual burden of obesity among ELA-affected SMW in their midlife. The study investigators developed an app-based MBI (28 daily modules, self-paced), "Eat Right Now" (ERN), which uses mindfulness to target craving-based eating.

The current single-arm, exploratory clinical trial evaluates the utility of ERN among mid-aged sexual minority women who are overweight (BMI larger or equal to 25) and have a history of early life adversities. Specifically, two aims guide the study: (1) Investigators will examine the feasibility and acceptability of ERN among mid-aged sexual minority women who are overweight and have a history of early life adversities. Exit-interviews will be conducted to understand women's experience and inform future adaptation of the intervention. (2) Preliminary, pre-post trial efficacy will be evaluated.

Participants will be screened using a two-part process taking place online, via an online screener and a Zoom-based screening. Research assessments will take place at baseline, post-intervention, and 4-month follow-up, digitally using using Qualtrics, LLC (Provo, UT, USA) survey management tool. Exit-interviews at post-intervention will be conducted via Zoom.

DETAILED DESCRIPTION:
Sexual minority women (SMW) in mid-age are at significantly higher risk for obesity, which is associated with greater vulnerability to cardiovascular disease, diabetes, cancer, and mortality. Further, this group also has elevated risk of early life adversities (ELA), such as childhood trauma and abuse. ELA has been linked to increased risks of midlife obesity and food addiction. However, interventions addressing this public health issue among SMW is scarce.

Mindfulness-based interventions (MBI), delivered via smartphone, could be an effective approach to reduce the dual burden of obesity among ELA-affected SMW in their midlife. Our team has developed an app-based MBI (28 daily modules, self-paced), known as "Eat Right Now" (ERN), which uses mindfulness to target craving-based eating. Results from a pilot study where ERN was administered to a general population of 64 adults showed promising results. However, despite these promising outcomes, no MBI, including ERN, has been tested specifically in ELA-affected adults including SMW. The potential effect of ERN as an MBI to enhance emotion regulation and mental health is also unknown.

Our team's overarching goal is to address the behavioral health burden of ELAs among SMW in midlife through mindfulness-based intervention and evaluate the biopsychosocial mechanisms of MBI for this population. The two (abbreviated) aims of this research study are: Aim 1. Examine the acceptability and preliminary efficacy of ERN as an internet-delivered MBI for distressed, overweight (BMI greater or equal to 25) ELA-affected SMW in midlife (age 30-54; n = 30). Aim 2. Investigate the mechanisms of ERN for ELA-affected SMW.

This is a stage 1 single arm trial where investigators hope to enroll 30 sexual minority women (SMW) aged 30-55, who meet all inclusion and exclusion criteria, including having a BMI>25, who are experiencing food cravings and endorsed overeating of these foods and who have experienced early life adversity (ELA).

Screening for eligibility will take place in a two-step process: (1) completion of a 5-10-minute online survey and (2) a face-to-face 15-25-minute zoom interview with a trained staff member. Given the online, remote nature of the study, a waiver of documentation of informed consent has been granted. Participants will be given a copy of the ICF at both screening steps. A trained research staff member will review all components of the ICF with the participant during the zoom interview.

Eligible participants will then be invited to complete an online baseline assessment designed to take up to one hour. Once complete, participants will be given access to the mobile-based mindfulness eating app and will be asked to complete it over the course of six to eight weeks.

Self-reported weight measurements will be taken periodically throughout the study using a standardized weight scale mailed to participants prior to the start of the intervention.

Participants that complete the self-paced intervention will then be invited to complete a 60-90-minute exit interview conducted via zoom with trained research staff. Online follow up assessments will also be conducted at 2-month and 4-month post-intervention.

ELIGIBILITY:
Inclusion Criteria: (a) 30-55 years of age; (b) BMI ≥ 25; (c) fluent in English; (d) have a smartphone; (e) reside in the U.S.; (f) experience food (salty or sweet) cravings and endorsed overeating of these foods (i.e. responded 'yes' to 'do you find yourself eating more than you'd like of a particular food or category of foods?') at least 4 times per week; (g) self-identify as a sexual minority woman (e.g., lesbian, bisexual, queer, or other sexual minority women); and (h) experienced early life adversity, screened via an adapted measure of childhood abuse.

Exclusion Criteria: (a) current eating disorder; (b) current strict diet (e.g. paleo, keto, vegan, calorie restriction); (c) current insulin use; (d) pregnant or trying to become pregnant; (e) previous use of the "Eat Right Now" application; and (f) history of serious mental illness, such as bipolar or psychotic disorders or self-injurious behaviors.

Ages: 30 Years to 55 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult
Gender Based: Yes — Female sex at birth
Enrollment: 30 (Actual)
Dates: Start 2021-11-02 (Actual); Primary Completion 2022-04-30 (Actual); Study Completion 2022-04-30 (Actual)

PRIMARY OUTCOMES:
Feasibility of ERN as measured by retention rates at 2-months | 2 months
  We will calculate rates of retention at post-intervention and 2-months follow-up as one of the feasibility outcomes.
Feasibility of ERN as measured by retention rates at 4-months | 4 months
  We will calculate rates of retention at post-intervention and 4-months follow-up as one of the feasibility outcomes.
Feasibility of ERN as measured by participation rates | 2 months
  We will calculate the rates of module completion by enrolled participants as an indicator of the feasibility of the program.
Acceptability of ERN as measured by the Client Satisfaction Questionnaire (CSQ) | 2 months
  The Client Satisfaction Questionnaire (CSQ) will assess participants' satisfaction with recruitment, retention, and intervention procedures. An overall score is produced by summing all item responses. For the CSQ-8 version, scores range from 8 to 32, with higher values indicating higher satisfaction.
Acceptability of ERN as measured by the adapted system usability scale | 2 months
  The system usability scale will assess acceptability of the app and various aspects of its usability.

SECONDARY OUTCOMES:
Food craving, assessed by Food Craving Questionnaire-Trait-Reduced (FCQ-Tr) at 2-months | 2 months
  The Food Craving Questionnaire-Trait-Reduced (FCQ-Tr) will assess participants' experience of food craving. Scores range from 15 to 75 with higher scores indicating higher levels of craving.
Food craving, assessed by Food Craving Questionnaire-Trait-Reduced (FCQ-Tr) at 4-months | 4 months
  The Food Craving Questionnaire-Trait-Reduced (FCQ-Tr) will assess participants' experience of food craving. Scores range from 15 to 75 with higher scores indicating higher levels of craving.
Reward-based eating, assessed by the Reward-based Eating Drive (RED) scale at 2-months | 2 months
  The Reward-based Eating Drive (RED) scale will assess participants' experience of reward-based eating. Overall scores range from 0 to 52 with higher scores indicating more engagement with reward-based eating.
Reward-based eating, assessed by the Reward-based Eating Drive (RED) scale at 4-months | 4 months
  The Reward-based Eating Drive (RED) scale will assess participants' experience of reward-based eating. Overall scores range from 0 to 52 with higher scores indicating more engagement with reward-based eating.
Mindfulness, assessed by the Five Facet Mindfulness Questionnaire (FFMQ) at 2-months | 2 months
  The Five Facet Mindfulness Questionnaire (FFMQ) will assess participants' self-reported mindfulness level. Total scores range from 39 to 195 with higher scores indicating greater levels of mindfulness. Sub-scale scores as well as mean scoring are also able to be obtained.
Mindfulness, assessed by the Five Facet Mindfulness Questionnaire (FFMQ) at 4-months | 4 months
  The Five Facet Mindfulness Questionnaire (FFMQ) will assess participants' self-reported mindfulness level. Total scores range from 39 to 195 with higher scores indicating greater levels of mindfulness. Sub-scale scores as well as mean scoring are also able to be obtained.
Mindfulness, assessed by the Mindful Awareness and Attention Scale (MAAS) at 2-months | 2 months
  The Mindful Awareness and Attention Scale (MAAS) will assess participants' self-reported mindfulness level. Scoring is obtained by computing a mean score for the 15-items. Scores range from 1 to 6 with higher scores reflecting greater levels of dispositional mindfulness.
Mindfulness, assessed by the Mindful Awareness and Attention Scale (MAAS) at 4-months | 4 months
  The Mindful Awareness and Attention Scale (MAAS) will assess participants' self-reported mindfulness level. Scoring is obtained by computing a mean score for the 15-items. Scores range from 1 to 6 with higher scores reflecting greater levels of dispositional mindfulness.
Depression, assessed by the Patient Health Questionnaire (PHQ-9) at 2-months | 2 months
  The Patient Health Questionnaire (PHQ-9) will assess participants' depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater severity of depression. Scale is self-report; responses should be verified by a clinician for true diagnosis of depression.
Depression, assessed by the Patient Health Questionnaire (PHQ-9) at 4-months | 4 months
  The Patient Health Questionnaire (PHQ-9) will assess participants' depressive symptoms. Scores range from 0 to 27, with higher scores indicating greater severity of depression. Scale is self-report; responses should be verified by a clinician for true diagnosis of depression.
Emotional regulation, assessed by the Difficulties in emotion regulation scale (DERS) at 2-months | 2 & 4 months
  The Difficulties in emotion regulation scale (DERS) short form is an 18-item scale that will assess participants' emotional regulation skills. Scores can be summed or averaged for interpretation. Total scores range from 18 to 90 with higher scores indicating greater emotion regulation.
Emotional regulation, assessed by the Difficulties in emotion regulation scale (DERS) at 4-months | 4 months
  The Difficulties in emotion regulation scale (DERS) short form is an 18-item scale that will assess participants' emotional regulation skills. Scores can be summed or averaged for interpretation. Total scores range from 18 to 90 with higher scores indicating greater emotion regulation.
Weight, measured by a standardized scale at 2-months | 2 months
  Change in weight and BMI will be assessed using a standardized scale provided to participants at baseline.
Weight, measured by a standardized scale at 3-months | 3 months
  Change in weight and BMI will be assessed using a standardized scale provided to participants at baseline.
Weight, measured by a standardized scale at 4-months | 4 months
  Change in weight and BMI will be assessed using a standardized scale provided to participants at baseline.

CONTACTS AND LOCATIONS:
Overall Officials: Shufang Sun, PhD, Principal Investigator — Brown University
Locations (1):
- Brown University, Providence, Rhode Island, United States

IPD SHARING:
Plan to Share IPD: Yes
External researchers interested in utilizing these data will be encouraged to do so provided they adhere to participant confidentiality requirements stipulated by the research study protection of human subjects protocol and the Brown University IRB.
Supporting Information: Study Protocol, ICF
Time Frame: Within 1.5 years of study completion.
Access Criteria: Please contact the principal investigator, Shufang Sun, PhD, at shufang_sun@brown.edu